CLINICAL TRIAL: NCT02833493
Title: Observational Study of MRI Monitoring in Patients With Aplastic Anemia (AA) and Low or Int-1 Risk of Myelodysplastic Syndromes(MDS) Complicated With Iron Overload
Brief Title: Study of MRI Monitoring in Patients With Aplastic Anemia and Low or Int-1 Risk of MDS Complicated With Iron Overload
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Bing Han, Department of Hematology, Peking Union Medical College Hospital
Other Study IDs: CICL670AAU05
Record Dates: First submitted 2016-07-05; First posted 2016-07-14 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Aplastic Anemia; Dysmyelopoietic Syndromes; Iron Overload
Keywords: Magnetic Resonance Imaging; Iron overload; Iron chelation therapy; Follow-up
MeSH Terms: conditions — Anemia, Aplastic; Myelodysplastic Syndromes; Iron Overload

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The investigators aim to give an overview of Iron overload(IOL) of patients with AA and low and int-1 risk MDS and their sequelae under different chelation treatment. And the investigators also aim to evaluate the relationship of LIC and T2*/R2*.

DETAILED DESCRIPTION:
Long-term transfusion therapy, a supporting treatment for patients with intractable chronic anemia is currently the most frequent cause of secondary iron overload. Both Aplastic anemia (AA) and low risk (low and intermediate-1 risk) myelodysplastic syndromes (MDS) are classified into bone marrow failure syndromes (BMFs) as they have a lot of characters in common. Iron overload (IOL) can then become a significant problem in regularly transfused patients, leading to organ damage, particularly in the liver and heart. Iron overload also has a suppressive effect on erythroid progenitors and may increase transfusion requirements. In those cases, iron chelation therapy may help to improve their quality of life and prolong their survival.

Because of the importance of iron chelation in patients with AA and low and intermediate-1(int-1) risk MDS complicated with iron overload, it is necessary to monitor their iron overload status to find the suitable patients to be chelated and follow up the effectiveness of therapy. Using quantitative Magnetic resonance imaging (MRI) T2* to detect the iron deposit of different organs has been introduce to China since 5 years ago. Compared to the traditional methods for evaluating iron overload like clinical manifestations, serum ferritin (SF) level, transferrin saturation (TS), CT and echocardiography (UCG) etc., which are widely used so far in China, MRI T2* provides an more accurate, convenient and affordable non-invasive way of monitoring iron overload. More important, it is very reliable to monitor the improvement of iron chelation therapy since the variation of MRI detection between different detections is very low. Few reports have been focused on IOL of MDS and AA in China so far.

Measurement of liver iron concentration (LIC) by MRI yields similar results to those coming from liver biopsy analysis, and is a validated tool for detection of iron overload. Data has been published from a multi-center trial evaluating the efficacy and safety of deferasirox (DFX) in low and intermediate-1 risk MDS patients with transfusion-dependent IOL and showed DFX yields sufficient reduction of excess iron indicated by serum ferritin levels and most importantly by liver MRI. But the median duration of DFX treatment is only 354 days and no data of Chinese patients was included. Most of the studies for MDS lack data of long term follow-up and there is scarcely any data on AA so far.

In China, more and more patients with iron overload can afford adequate iron chelation therapies, although there are still some patients who cannot afford at all or can only be chelated irregularly. And some patients can only accept deferoxamine instead of deferasirox because of the medical insurance policies. It is important to include patients with different situations and monitor their iron change in their major organs based on different chelation level.

In this study, it is anticipated to evaluate prospectively 80 patients with AA and low or int-1 risk MDS with IOL, by the traditional methods and MRI T2*. Clinical parameters and T2*values will be monitored every 12 months for 3 years. Other parameters like clinical follow-ups ( rate of infection, liver disease, cardiac disorders, endocrine function and other co-morbidities associated with MDS/AAs, etc.), SF, liver and kidney function, UCG tests will be monitored as well at the interval of every 6 months. At the end of the study, patients will be classified as well chelated groups (defined as those received deferasirox 20mg/kg or deferoxamine 40 mg/kg for more than 255 days/year) or poor chelated groups (defined as those received iron chelation therapy dose less than above) and compared the differences of their outcome and change of iron status. The investigators aim to give an overview of IOL of patients with AA and low and int-1 risk MDS and their sequelae under different chelation treatment. And the investigators also aim to evaluate the relationship of LIC and T2*/R2*. It is the first and longest prospective clinical trial on AA and low risk MDS and will give us a better understanding of the value of proper chelation treatment for the organ function.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of 18-80 year old.
2. With blood transfusion history or RBC-transfusion-dependence.
3. BM smear and biopsy plus chromosome analysis within 3 months before signing ICF, otherwise done during screening.
4. Excluding other diseases which might cause hematological abnormalities.
5. Serum ferritin level≥500ng/ml with no sign of active infection or malignant disease.
6. Treatment with underlying disease is permitted for non-hematological and hematological conditions.
7. Previous iron chelation therapy like deferasirox or deferoxamine is permitted.
8. ECOG performance score ≤2
9. All subjects must: agree not to donate blood or be counseled about pregnancy precautions and risks of fetal exposure.
10. Written informed consent.

Exclusion Criteria:

1. Patients who are under 18-year-old or over 80-year-old.
2. Prior history of other cancer unless cancer-free for ≥5 years.

   Subjects with the following history/concurrent conditions may enroll at any time:

   Basal cell carcinoma of the skin Squamous cell carcinoma of the skin Prostate cancer stage-1
3. Proved HIV-1 infection
4. Active HBV or active HCV infection.
5. Pregnant or lactating
6. Patients unwilling to or unable to comply with the protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AA or MDS with very good, good and intermediate risk as per IPSS-R who meet all the following criteria.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-09 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
MRI T2*/R2* for liver and heart | 3 years

IPD SHARING:
Plan to Share IPD: Undecided